CLINICAL TRIAL: NCT05489380
Title: Optical Diagnosis Versus Laser Measurement of Polyps' Size During Colonoscopy and Implications for Surveillance (Polyp Size Study)
Brief Title: Optical Diagnosis Versus Laser Measurement of Polyps' Size During Colonoscopy and Implications for Surveillance
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government); Erasmus Medical Center (Other); Bnai Zion Medical Center (Other Government); NYU Langone Health (Other); Indiana University Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: NL80961.091.22
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Polyp
Keywords: screening; colonoscopy; surveillance

STUDY DESIGN:
Intervention Model Description: As optical assessment of polyps has a high interobserver variability, the order of polyps' size measurement using biopsy forceps or AM will be randomized per patient. Therefore, this study consists of two arms: Optical polyp size assessment, followed by biopsy forceps and then AM measurement (1), and optical assessment, followed by AM measurement and then biopsy forceps assisted assessment (2) (Figure 1).
Who Masked: Outcomes Assessor
Masking Description: the endoscopist will remain blinded to the AccuMeasure measurement outcomes, to avoid a learning effect that could influence subsequent measurements. Even so, all pathologist assessments will be done independent of the study allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Accumeasure last (Other): Optical polyp size assessment, followed by biopsy forceps and then AccuMeasure measurement
  Interventions: Device: AccuMeasure
- AccuMeasure first (Other): optical assessment, followed by AccuMeasure measurement and then biopsy forceps assisted assessment (2)
  Interventions: Device: AccuMeasure

INTERVENTIONS:
Device: AccuMeasure — intracolonoscopy measurement of polyps using a laser-based device
  Other Names: laser-based polyp measurement

SUMMARY:
Recent updates of the guidelines on polyp surveillance of the American Society of Gastrointestinal Endoscopy (ASGE) and European Society of Gastrointestinal Endoscopy (ESGE) increasingly focus on size of polyps as an important indicator of malignant transformation to colorectal cancer (CRC). However, the interobserver variability in polyp size assessment between optical diagnosis of endoscopists and pathologists is considerable. This may lead to incorrect surveillance intervals in patients at risk for developing colorectal cancer, which may increase the risk of post-colonoscopy CRC (PCCRC). This study aims to assess the precision of a new laser-based measurement system (AccuMeasure, VTM Technologies Ltd.) for polyps during colonoscopy.

DETAILED DESCRIPTION:
Objective: The main objective is to compare the precision of polyp size measurement by AccuMeasure to biopsy forceps assisted measurement. Secondary objectives are to assess: Time needed for measurement and learning curve, endoscopists advised surveillance intervals based on both measurement methods, and safety.

Study design: Multicenter, randomized, parallel group, endoscopist blinded study, including the measurement of 138 polyps during standard colonoscopy. With a polyp detection rate of approximately 40%1, this results in up to 345 patients/colonoscopies to be included. Enrollment will conclude once 138 polyps are included in the study.

Study population: All adult patients with screening or surveillance colonoscopies will be asked for informed consent. Polyps smaller than 25mm found during colonoscopy are considered eligible for inclusion. Up to 3 polyps per patient can be included in this study.

Intervention: Optical assessment will be performed upon identification of the polyp. Then, measurement with AccuMeasure and biopsy forceps will be performed in a randomized order. The endoscopist will remain blinded to the AccuMeasure measurement outcomes, to avoid a learning effect that could influence subsequent measurements.

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients (>18 years)

  * Scheduled for screening, surveillance, or diagnostic colonoscopy
  * Polyps of all forms ≤ 25mm as assessed by the endoscopist

Exclusion Criteria:

* • Therapeutic colonoscopy;

  * Inflammatory bowel disease (IBD);
  * American Society of Anesthesiologists (ASA) score of >3;
  * Inadequately corrected anticoagulation disorder or anticoagulation medication use;
  * Inability to provide informed consent;
  * Inadequate bowel preparation (Boston bowel preparation scale score [BBPS] <2 per segment);
  * No polyps identified during colonoscopy or only small (<5mm) hyperplastic rectal polyps;
  * Intraprocedural complications, not caused by the study device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Cohens' Kappa coefficient | at colonoscopy
  interobserver agreement between AccuMeasure and biopsy forceps assisted measurement

SECONDARY OUTCOMES:
Number of Participants with adverse events up to 30 days post colonoscopy | 30 days post colonoscopy
  Number of Participants with adverse events
Absolute size differences | at colonoscopy
  Size differences for optical/biopsy forceps/AM assessment as compared to pathology size measurement;
Time for measurement | at colonoscopy
  Time for measurement with AccuMeasure related to number of measurements performed
Endoscopist advised surveillance interval | At colonoscopy
  Endoscopist advised surveillance interval based on optical assessment during colonoscopy, on measurement with an open biopsy forceps, and on measurement with AccuMeasure

OTHER OUTCOMES:
Method of polyp removal | at colonscopy
  method of polyp removal, i.e., polypectomy, endoscopic mucosal resection, endoscopic submucosal dissection
BBPS | at colonoscopy
  Boston bowel preparation scale score (BBPS), in which segmental scores of 0 are worst and scores of 3 are best (completely clean)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Indiana University Hospital, Indianapolis, Indiana
  - NYU Langone Health, New York, New York
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The dataset used during this study is available from the corresponding author upon reasonable request
Supporting Information: SAP, CSR, Analytic Code
Time Frame: 15y
Access Criteria: The dataset used during this study is available from the corresponding author upon reasonable request